CLINICAL TRIAL: NCT00910663
Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalence Study of Mycophenolate Mofetil Capsules Under Fed Conditions
Brief Title: Mycophenolate Mofetil 250 mg Capsules Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-983-AU
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (mycophenolate mofetil) First (Experimental): Mycophenolate Mofetil 250 mg Capsule dosed in first period followed by Cellcept® 250 mg Capsule dosed in second period.
  Interventions: Drug: Mycophenolate Mofetil
- Reference (CellCept®) First (Active Comparator): CellCept® 250 mg Capsule dosed in first period followed by Mycophenolate Mofetil 250 mg Capsule dosed in second period.
  Interventions: Drug: CellCept®

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 250 mg Capsule
  Arms: Test (mycophenolate mofetil) First
Drug: CellCept® — 250 mg Capsule
  Arms: Reference (CellCept®) First

SUMMARY:
The objective of this study was to compare the oral availability of a test product of Mycophenolate Mofetil 250 mg capsule to an equivalent oral dose of the commercially available reference product, CellCept® 250 mg capsule administered to healthy subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria to be considered for study participation:

* Subject must be male or non-pregnant, non-breast-feeding female
* Subject must be at least 18 years of age
* Subject must have a Body Mass Index (BMI) between 19 and 30 kg/m2, inclusive, and body weight should be at least 50 kg (110 lbs)
* Female Subjects - not surgically sterile or at least two years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, double barrier (condom with spermicide, diaphragm with spermicide), intra-uterine device (IUD), or vasectomized partner (6 months minimum since vasectomy).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to the start of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period and return for any outpatient visits.

Exclusion Criteria:

Subjects may be excluded for any of the following:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition which, in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG or clinical laboratory results at screening.
* History or presence of allergic or adverse response to mycophenolate mofetil or related drugs.
* Has been on a significantly abnormal diet during the four weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, including hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Has been treated with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 90 days prior to the first dose of study medication.
* Is a female with a positive pregnancy test result.
* Female who has used implanted hormonal contraceptives anytime during the 6 months prior to study start.
* Has an intolerance to venipuncture.
* Has difficulty fasting or consuming standard meals.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates)
* Has a history of drug or alcohol abuse.
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Bieberdorf, MD, Principal Investigator — Cedra Clinical Research, LLC
Locations (1):
- Cedra Clinical Research, LLC, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil (Test) First: Mycophenolate Mofetil 250 mg Capsule dosed in first period followed by Cellcept® 250 mg Capsule dosed in second period.
- CellCept® (Reference) First: CellCept® 250 mg Capsule dosed in first period followed by Mycophenolate Mofetil 250 mg Capsule dosed in second period.
Period: Period 1
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 18 | 12 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 22 | 18 | 40
  Black | 3 | 8 | 11
  Asian | 0 | 1 | 1
  American Indian | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Bioequivalence based on Cmax - Maximum Drug Concentration
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Mycophenolate Mofetil (Test): Mycophenolate Mofetil 250 mg Capsule dosed in either period
- CellCept® (Reference): CellCept® 250 mg Capsule dosed in either period.
Arm/Group | Mycophenolate Mofetil (Test) | CellCept® (Reference)
Number analyzed (Participants) | 59 | 59
µg/mL | 2.8358 (0.9056) | 2.9768 (1.2500)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil (Test) vs CellCept® (Reference); Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 97.01, 90% CI [90.01 to 104.55] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf
Description: Bioequivalence based on AUC0-inf - Area under concentration-time curve from time zero to infinity (extrapolated)
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Mycophenolate Mofetil (Test) | CellCept® (Reference)
Number analyzed (Participants) | 59 | 59
µg*h/mL | 14.6569 (3.8700) | 14.2048 (3.9281)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil (Test) vs CellCept® (Reference); Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 102.81, 90% CI [100.23 to 105.45] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t
Description: Bioequivalence based on AUC0-t - Area under concentration-time curve from time zero to time of last non-zero concentration
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Mycophenolate Mofetil (Test) | CellCept® (Reference)
Number analyzed (Participants) | 59 | 59
µg*h/mL | 13.8388 (3.7728) | 13.4016 (3.8398)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil (Test) vs CellCept® (Reference); Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 103.35, 90% CI [100.51 to 106.27] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

ADVERSE EVENTS:
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 6/60 | 1/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (Test) First (N=60) | CellCept® (Reference) First (N=60)
Headache (Vascular disorders) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is not permitted to discuss or publish trial results.